CLINICAL TRIAL: NCT07062042
Title: Styrkende Narrativ: Hjelp Til Selvhjelp for Ukrainske Flyktninger / Empowering Narratives: Help to Self-help to Ukrainian Refugees
Brief Title: Empowering Narratives
Acronym: EN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kristiania University College (Other)
Collaborators: University of Konstanz (Other); Oswaldo Cruz Foundation (Other); Mental helse (Unknown); Vårsta Diakoni (Unknown); Norsk-Ukrainsk hjelpeorganisasjon (Unknown); The Dam Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Styrkende Narrativ Kristiania; 547119 (Other Grant/Funding Number: Stiftelsen DAM)
Record Dates: First submitted 2025-06-10; First posted 2025-07-14 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: PTSD - Post Traumatic Stress Disorder; Depression Disorders; Dissociation; Refugee
Keywords: PTSD; Depression Disorders; Dissociation; Ukrainian Refugees; Norway; Narrative Exposure Therapy
MeSH Terms: conditions — Combat Disorders; Dissociative Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This study utilizes a parallel-group randomized controlled trial design. Participants will be randomly assigned to one of two groups: an intervention group, which will receive Narrative Exposure Therapy (NET), and a waitlist control group, which will receive treatment after the initial study period (when the post-treatment screening of the participant that is matching case for each control case is concluded).
  Quantitative data will be collected from both groups using a repeated screening measures approach. For the intervention group, data will be gathered at three timepoints: (1) baseline (prior to treatment), (2) post-treatment (approximately one week after the final session), and (3) follow-up (six months after treatment completion). For the control group, data will be collected at two timepoints: (1) baseline, and (2) after a waiting period equivalent in length to the intervention group's treatment phase, prior to their own treatment onset.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case (Experimental): Participants assigned to that arm receive Narrative Exposure Therapy (intervention) immediately after the baseline screening
  Interventions: Behavioral: Narrative Exposure Therapy
- Control (No Intervention): Waiting List: the participant waits and receives no intervention until the treatment and the re-screening of the case participant is done. Then the control participant, assigned to the waiting list, receive the same intervention.

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy — Narrative Exposure Therapy (NET) is a short-term, trauma-focused intervention developed for individuals exposed to multiple traumatic events, including refugees and survivors of war and organized violence. It is grounded in principles of cognitive-behavioral therapy and testimonial therapy. NET helps adults reconstruct a coherent narrative of their life by integrating fragmented traumatic memories through structured exposure within a chronological autobiographical framework. Core components include lifeline construction, imaginal exposure to traumatic events, and reprocessing of emotional responses. The method emphasizes stabilization through therapeutic structure and is supported by evidence from randomized controlled trials showing reductions in PTSD symptoms. The approach is protocol-driven and applicable in low-resource settings under supervision, as outlined in the practice document.
  Arms: Case

SUMMARY:
Background: The Russian invasion of Ukraine has resulted in forced displacement, with over 80,000 Ukrainian refugees now residing in Norway. This displacement has led to increased vulnerability to trauma and mental health challenges. Narrative Exposure Therapy (NET), a short-term trauma-focused intervention, has demonstrated efficacy in reducing PTSD symptoms among individuals exposed to organized violence and war.

Aim: The protocol aims to assess the clinical effects of Narrative Exposure Therapy (NET) on PTSD and depression symptoms among Ukrainian refugees in Norway and to facilitate training and supervised practice for Ukrainian health professionals and workers in using NET.

Methods: This study employs a pretest-posttest randomized controlled experimental design. Ukrainian health professionals and workers in Norway will receive standardized NET training through a digital course. Subsequently, they will treat Ukrainian refugees using NET under supervision. Participants will be screened and assessed at three time points: baseline, immediately after treatment, and at 6-month follow-up. Validated questionnaires in Ukrainian and Russian will be used: PHQ-9, ITQ, LEC-5, SHUT-D, and demographic questionnaire. Exclusion criteria include active psychotic spectrum disorders, neurodevelopmental disorders and concurrent trauma therapy.

DETAILED DESCRIPTION:
Ethical Approval:

The study received ethical approval from the Regional Committees for Medical and Health Research Ethics - South-East D (REK sør-øst D) in Norway, under reference number 790305.

Quality Assurance and Data Management:

The proposed study will not use any registry data and instead collect data with validated questionnaires. Questionnaires will be filled in during interviews with the NET therapist, which will increase data quality by ensuring that participants understand the questions and are engaged in answering them. The questionnaires were translated to Ukrainian by the Trauma Consortium, which helps to ensure both quality and understanding from both patients and health workers. Questionnaire data will be coded in accordance with the published manuals for the respective questionnaires, and a data dictionary will be used to describe each variable according to the manuals.

All data, including notes from NET sessions and the resulting narratives, will be stored on a secure server, TSD (link to the website can be found in the reference list). Questionnaire data will be collected with a secure and anonymous data collection tool, Nettskjema (link to the website can be found in the reference list), and will be directly transferred to TSD. The study will also include a link key, stored in TSD, that links the participant's name to an anonymous code, and the anonymous code to the dataset, so that data will not be stored together with the participants' names. The data management in the current study has been assessed with a Data Protection Impact Assessment (DPIA) and has been approved by the Norwegian Agency for Shared Services in Education and Research, SIKT (link to the website in the reference list) and the Norwegian Regional Committee for Medical and Health Research Ethics, REK (link to the website can be found in the reference list).

REK also approved an emergency procedure for handling cases where participants score highly on depression or suicidal thoughts. The procedure includes a psychoeducative conversation with the participants by the project's PI (Vanessa Nolasco Ferreira) and the offer to send a letter to the participant's General Practitioner, with information about the depression and/or suicidal thoughts score. This letter will allow the GP to refer the participant to the specialized mental health services and reduce waiting times for treatment.

Sample Size Assessment:

A convenience sampling approach will be utilized, with the final sample size depending on the number of individuals who volunteer and meet the inclusion criteria. This approach accommodates variability in participant availability and willingness. The project has financial resources for NET training of 25 health workers, and each health worker needs to conduct supervised NET with two participants as part of the practical training that is necessary for NET certification. We are therefore aiming at 50 participants (25 in the intervention group and 25 in the waitlist control group). Previous NET interventions in similar populations have shown significant effects with comparable or considerably smaller sample sizes.

Plan for Missing Data:

The dropout rate during NET interventions tends to be low or zero, partially due to the short duration of interventions. Therefore, we expect minimal risk of missing datasets at post-treatment assessments. There might be a slightly higher risk for missing datasets at 6-months follow-up. We will compare demographic data and initial post-treatment effects of any dropouts with data of participants that complete the follow-up assessment, in order to evaluate potential biases due to systematic differences between dropouts and completers. There is no risk of missing data due to incomplete questionnaires (i.e. participants accidentally not answering single items) since the software used for assessment does not allow submission of the questionnaire unless all items are answered.

ELIGIBILITY:
Inclusion Criteria:

* Ukrainian refugee residing in Norway.
* Arrival in Norway after 24 February 2022.
* Minimum 18 years old
* Provided informed consent for participation.
* Classified as having PTSD symptoms (ITQ) OR reported traumatic experience (LEC-5) OR present PTSD comorbidities (PHQ-9, Shut-D).

Exclusion Criteria:

* Diagnosis, history, or scores compatible with the psychotic spectrum
* Diagnostic of neurodevelopmental disorders
* Current participation in ongoing trauma-focused psychological treatment (e.g., therapy for PTSD).
* Declining consent for mandatory elements of the study (e.g., participation in screening or treatment delivery).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
PTSD Symptom Severity (ITQ) | Baseline, Post-treatment (one to seven days after the last treatment session), 6-month Follow-up (counted after the post-treatment screening)
  Assesses symptoms of PTSD and Complex PTSD, including re-experiencing, avoidance, threat perception, and functional impairment.
  Instrument: International Trauma Questionnaire (ITQ)
  Outcome Focus: Change in PTSD symptom scores over time (H1, H4)
Dissociation Symptoms (Shut-D) | Baseline, Post-treatment (one to seven days after the last treatment session), 6-month Follow-up (counted after the post-treatment screening)
  Measures dissociative responses specific to trauma, including cognitive-emotional shutdown, sensory-motor dissociation, and behavioral shutdown.
  Instrument: Shutdown Dissociation Scale (Shut-D)
  Outcome Focus: Change in dissociation symptom scores over time (H2, H5)
Depression Symptoms (PHQ-9) | Baseline, Post-treatment (one to seven days after the last treatment session), 6-month Follow-up (counted after the post-treatment screening)
  Measures the frequency of depressive symptoms over the past two weeks, including somatic and cognitive-affective dimensions, plus functional impairment.
  Instrument: Patient Health Questionnaire-9 (PHQ-9)
  Outcome Focus: Change in depressive symptoms (H3, H6)

SECONDARY OUTCOMES:
Exposure to Traumatic Events (LEC-5) | Baseline
  Captures direct and indirect exposure to 17 categories of potentially traumatic events, including whether the event "happened to me."
  Instrument: Life Events Checklist for DSM-5 (LEC-5)
  Association between level of trauma exposure and symptom severity (H7)

OTHER OUTCOMES:
Age | Baseline
  Age in years
Gender | Baseline
  Male, Female
Marital status | Baseline
  Single, have never been married; Married/co-habiting; Divorced/separated - within last year; Divorced/separated - for more than 1 year; Widow/Widower - within last year; Widow/Widower - for more than 1 year.
  Analytical Use: Covariates or moderators in outcome models
Education | Baseline
  Primary (less than 7 grades); Incomplete secondary (less than 10 grades); Trade factory apprenticeship or professional courses after 7-8 grades; Completed secondary (10-11 grades); Trade factory apprenticeship or professional courses after 10-11 grades; Secondary technical education; Uncompleted higher education (3 courses or less); Completed higher education.
  Instrument: Custom questionnaire
  Analytical Use: Covariates or moderators in outcome models
Long-term illness, health problem or handicap | Baseline
  Yes or No
General Perception of Health | Baseline
  Very good; Good ; Fair; Poor; Very poor.
Time in Norway | Baseline
  Patient reports during the first therapy session (lifeline session)
Functional Impairment | Baseline, Post-treatment (one to seven days after the last treatment session), 6-month Follow-up (counted after the post-treatment screening)
  In the international trauma questionaire function impairment connected to PTSD is measured if At least one of P7, P8, or P9 > 2 meets criteria for PTSD functional impairment (PTSDFI) If the patient meets the criteria for CPTSD the function impairment is measured if at least one of C7, C8, or C9 > 2 meets criteria for DSO functional impairment (DSOFI) In what concerns depression, the measure will come from the question number 10 in PHQ9 if the patient answers somewhat difficult, difficult or very difficult.
  Embedded in: ITQ and PHQ-9
  Outcome Focus: Supplementary analysis of clinical relevance

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Nolasco Ferreira, Associate Professor, PhD, Principal Investigator — Kristiania University of Applied Sciences
Locations (1):
- Kristinia University of Applied Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided
This study does not plan to share individual participant data (IPD) publicly. However, de-identified group-level results and relevant statistical outputs will be shared through peer-reviewed publication. A full study protocol will be submitted for peer review to the European Journal of Psychotraumatology, which adheres to ICMJE trial registration and transparency standards. The manuscript includes detailed methodological information, including hypotheses, intervention structure, outcome measures, and ethical safeguards. Upon publication, the protocol will be publicly accessible and cited in connection with the trial results.

REFERENCES:
- [Background] Schauer M, Neuner F, Elbert T. Narrative Exposure Therapy (NET) For Survivors of Traumatic Stress. 3 ed: Hogrefe Publishing; 2025
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Cloitre M, Shevlin M, Brewin CR, Bisson JI, Roberts NP, Maercker A, Karatzias T, Hyland P. The International Trauma Questionnaire: development of a self-report measure of ICD-11 PTSD and complex PTSD. Acta Psychiatr Scand. 2018 Dec;138(6):536-546. doi: 10.1111/acps.12956. Epub 2018 Sep 3. PMID 30178492
- [Background] Gray MJ, Litz BT, Hsu JL, Lombardo TW. Psychometric properties of the life events checklist. Assessment. 2004 Dec;11(4):330-41. doi: 10.1177/1073191104269954. PMID 15486169
- [Background] Schalinski I, Schauer M, Elbert T. The shutdown dissociation scale (shut-d). Eur J Psychotraumatol. 2015 May 13;6:25652. doi: 10.3402/ejpt.v6.25652. eCollection 2015. PMID 25976478
- [Background] Labberton AS, Ozeryansky L, Helland Y, Skogheim TS, Hansen TM. Trends in the health status of Ukrainian refugees in Norway according to month of arrival during 2022. BMC Public Health. 2024 Nov 12;24(1):3127. doi: 10.1186/s12889-024-20660-0. PMID 39533254
- [Background] Labberton AS, Hansen TM, Skogheim TS, Helland Y. Healthcare needs among refugees from Ukraine arriving in Norway during 2022. Norwegian Institute of Public Health; 2023 May 2023.
- [Background] Ardino V, Schalinski I. Recent developments of narrative exposure therapy. Maltrattamento e Abuso All'Infanzia: Rivista Interdisciplinare. 2020;.22(3):pp
- [Background] Tracy SJ. A phronetic iterative approach to data analysis in qualitative research. 질적연구. 2018;19(2):61-76
- [Background] Lely JCG, Smid GE, Jongedijk RA, W Knipscheer J, Kleber RJ. The effectiveness of narrative exposure therapy: a review, meta-analysis and meta-regression analysis. Eur J Psychotraumatol. 2019 Mar 25;10(1):1550344. doi: 10.1080/20008198.2018.1550344. eCollection 2019. PMID 31007868
- [Background] Wei Y, Chen S. Narrative exposure therapy for posttraumatic stress disorder: A meta-analysis of randomized controlled trials. Psychol Trauma. 2021 Nov;13(8):877-884. doi: 10.1037/tra0000922. Epub 2021 Feb 22. PMID 33617284
- [Derived] Ferreira VN, Hjelmervik H, Bell-Mizori AR, Tokovska M, Domogalla SA, Serpeloni F, Axelson S, Arango I, Weber S. Empowering narratives: aid to self-help for Ukrainian refugees: a randomized controlled trial of Narrative Exposure Therapy (NET) delivered by supervised Ukrainian health workers in Norway. Eur J Psychotraumatol. 2025 Dec;16(1):2567094. doi: 10.1080/20008066.2025.2567094. Epub 2025 Oct 27. PMID 41143444
- See also: UNHCR. The Operational Data Portal 2025 — https://data.unhcr.org/en/situations/ukraine
- See also: TSD, Tjenester for Sensitive Data - secure data storage server — https://www.uio.no/tjenester/it/forskning/sensitiv/
- See also: Nettskjema - secure questionnaire data collection tool — https://www.uio.no/tjenester/it/adm-app/nettskjema/
- See also: SIKT - Norwegian Agency for Shared Services in Education and Research — https://sikt.no/en/home
- See also: REK - Norwegian Regional Committee for Medical and Health Research Ethics — https://rekportalen.no/en/

DOCUMENTS (3):
  • Study Protocol: Ethical Committee (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT07062042/Prot_001.pdf
  • Study Protocol and Statistical Analysis Plan: Methods and Analysis (2025-08-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT07062042/Prot_SAP_003.pdf
  • Informed Consent Form (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT07062042/ICF_002.pdf